CLINICAL TRIAL: NCT06050577
Title: The Effect of Oral Semaglutide on Bone Turnover in Patients With Type 2 Diabetes: a Randomized Placebo-controlled Clinical Trial - (SOBER II)
Brief Title: The Effect of Oral Semaglutide on Bone Turnover in Patients With T2D: a Randomized Placebo-controlled Clinical Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EU CT: 2023-505959-45-00
Record Dates: First submitted 2023-09-08; First posted 2023-09-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes; Osteopenia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Bone Diseases, Metabolic | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oral Semaglutide/Rybelsus (Experimental): oral Semaglutide 7-14 mg (or highest tolerated dose) once daily for 52 weeks (incl. titration)
  Interventions: Drug: oral Semaglutide/Rybelsus
- oral Placebo (Placebo Comparator): oral Placebo 7-14 mg (or highest tolerated dose) once daily for 52 weeks (incl. titration)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: oral Semaglutide/Rybelsus — Weeks 1-4: 3 mg of oral semaglutide once daily. Weeks 5-52: 7 mg of semaglutide once daily as maintenance dose. Dose may be increased to 14 mg of semaglutide once daily as maintenance dose after 2 months if glucose levels are out of range.
  Arms: oral Semaglutide/Rybelsus
Drug: Placebo — Weeks 1-4: 3 mg of oral placebo once daily. Weeks 5-52: 7 mg of placebo once daily as maintenance dose. Dose may be increased to 14 mg of placebo once daily as maintenance dose after 2 months if glucose levels are out of range.
  Arms: oral Placebo

SUMMARY:
The hypothesis for this study is that oral Semaglutide, a GLP-1Ra, has a positive effect on the balance between build-up and degradation as well as the strength of the bones in men and women aged 50-85 years with type 2 diabetes and an increased risk of bone fractures. Treatment involves once daily oral GLP-1Ra semaglutide or matching placebo for 52 weeks. The effect will be measured by bone markers in blood samples, bone scans, bone tissue and bone marrow tests (bone marrow aspiration and biopsy), physical activity assessed by a questionnaire, and direct bone strength measured by microindentation at the start and end of the study.

ELIGIBILITY:
Inclusion criteria

* Type 2 diabetes and glycosylated haemoglobin (HbA1C) of 48-91 mmol/mol (6.5-10.5%) and
* T-score <-1 in hip or lower back, assessed by DXA scan and / or
* Low-energy fracture within the last 3 years

Exclusion criteria

* T-score <-2.5 in hip or lower back, assessed by DXA scan, although these individuals may be included if they are not candidates for conventional osteoporosis therapy, e.g., due to allergies and renal impairment, or if they prefer to participate in the trial.
* Type 1 diabetes mellitus
* Severe NPDR (non-proliferative diabetic retinopathy) or PDR (proliferative diabetic retinopathy) assessed within the last year. If a recent assessment is unavailable, a new retinal photo test will be performed.
* Congestive heart failure (NYHA Class IV)
* Primary hyperparathyroidism
* Vitamin D deficiency (<25 nM) (re-test after substitution acceptable)
* Known disorders affecting bone metabolism, e.g., uncontrolled thyrotoxicosis, severe renal impairment (eGFR <30) or liver dysfunction (baseline phosphatase higher than twice upper limit (105 U/L)), rheumatism, celiac disease, hypogonadism, severe COPD, hypopituitarism, Cushing's disease
* Clinically significant concomitant diseases or disorders (e.g., cancer) or clinically significant abnormal values in laboratory screening tests, including increased Choriogonadotropin (hCG) in women.
* History of gastrointestinal surgery (except uncomplicated surgical procedures such as hernia surgery and appendectomy)
* Antiresorptive or bone anabolic drugs for the last 12 months
* Use of anabolic steroids in the previous year
* Use of GLP-1Ras within 90 days
* Stable therapy with DPP4 inhibitors (unless the patient is willing to discontinue the treatment)
* History of pancreatitis
* Allergy or hypersensitivity to the active substance or to any of the ingredients
* Inability to give informed consent
* Previous bariatric surgery
* BMI <20 kg/m2 or BMI>37 kg/m2

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Procollagen type 1 N-terminal propeptide (P1NP) | Baseline and 52 weeks
  Percentage changes in bone formation marker P1NP from baseline and after 12 months

SECONDARY OUTCOMES:
Collagen 1 cross link C-terminal telopeptide (CTX) | Baseline and 52 weeks
  Changes in bone resorption marker CTX from baseline and after 12 months
Osteocalcin | Baseline and 52 weeks
  Changes in bone formation marker osteocalcin from baseline and after 12 months
Bone specific alkaline phosphatase (BALP) | Baseline and 52 weeks
  Changes in bone formation marker BALP from baseline and after 12 months
Bone mineral density (BMD) | Baseline and 52 weeks
  Changes in BMD (total hip, femoral neck and lumbar spine (L1-4)) assessed by DXA scans from baseline and after 12 months
Estimated bone strength | Baseline and 52 weeks
  Changes in estimated bone strength assessed by finite elemental analysis (HR-pQCT scan) from baseline and after 12 months
Total volumetric BMD | Baseline and 52 weeks
  Changes in total volumetric BMD (mg/cm^3) assessed by HR-pQCT scan of distal tibia and radius
Trabecular volumetric BMD | Baseline and 52 weeks
  Changes in trabecular volumetric BMD (mg/cm^3) assessed by HR-pQCT scan of distal tibia and radius
Cortical volumetric BMD | Baseline and 52 weeks
  Changes in cortical volumetric BMD (mg/cm^3) assessed by HR-pQCT scan of distal tibia and radius
Bone volume | Baseline and 52 weeks
  Changes in trabecular bone volume pr total volume (BV/TV) assessed by HR-pQCT scan of distal tibia and radius
Trabecular thickness | Baseline and 52 weeks
  Changes in trabecular thickness (mm) assessed by HR-pQCT scan of distal tibia and radius
Cortical thickness | Baseline and 52 weeks
  Changes in cortical thickness (mm) assessed by HR-pQCT scan of distal tibia and radius
Cortical porosity | Baseline and 52 weeks
  Changes in cortical porosity assessed by HR-pQCT scan of tibia and radius
Bone formation rate | 52 weeks
  Changes in bone formation rate (BRF/BS, µm^3/µm^2 per day), the volume of mineralized bone made per unit surface of bone per year, based on dynamic histomorphometry of bone tissue
Fat tissue distribution | Baseline and 52 weeks
  Change in fat tissue distribution, assessed by DXA
Lean tissue distribution | Baseline and 52 weeks
  Change in lean tissue distribution, assessed by DXA
Glycosylated haemoglobin (HbA1C) | Baseline and 52 weeks
  Change in HbA1c from baseline and after 12 months
Physical activity | Baseline and 52 weeks
  Change in physical activity based on analysis of International Physical Activity Questionnaire Short Form (IPAQ-SF) from baseline and after 12 months
Body mass index (BMI) | Baseline and 52 weeks
  Change in BMI from baseline and after 12 months

OTHER OUTCOMES:
Osteogenic potential | 52 weeks
  Change in osteogenic potential, i.e., ability to form new bone, assessed using spatial transcriptomics and single-cell RNA sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No